CLINICAL TRIAL: NCT00867165
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Efficacy and Safety Study of Ezetimibe Monotherapy in Children (Ages 6 to 10 Years) With Primary Hypercholesterolemia (Heterozygous Familial and Nonfamilial) (Phase 3, Protocol No. P05522)
Brief Title: Pediatric Study to Evaluate the Efficacy and Safety of Ezetimibe Monotherapy in Children With Primary Hypercholesterolemia (P05522)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05522; 2008-006271-70 (EudraCT Number); MK-0653-170 (Other: Merck Study Number)
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Results first posted 2013-05-30 (Estimated); Last update posted 2024-05-21 (Actual); Status verified 2022-02

CONDITIONS: Primary Hypercholesterolemia
Keywords: heterozygous familial hypercholesterolemia; nonfamilial hypercholesterolemia
MeSH Terms: interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ezetimibe (Experimental): Ezetimibe 10-mg tablet once daily for 12 weeks
  Interventions: Drug: ezetimibe
- Placebo (Placebo Comparator): Placebo to match ezetimibe 10-mg tablet once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ezetimibe — oral tablets: ezetimibe 10 mg once daily for 12 weeks
  Other Names: SCH 58235; MK-0653; Zetia
  Arms: Ezetimibe
Drug: Placebo — oral tablets: placebo to match ezetimibe 10 mg; administered once daily during the 5-week, single-blind, placebo run-in and diet stabilization period and 12-week double-blind treatment period
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of ezetimibe 10 mg/day compared to placebo on the reduction of low-density lipoprotein cholesterol (LDL-C) from baseline to 12 weeks of treatment in children >=6 to <=10 years old with primary hypercholesterolemia. The study will also evaluate the effect of ezetimibe on total cholesterol (TC), apolipoprotein B (Apo B), high-density lipoprotein cholesterol (HDL-C), non-HDL-C, and triglycerides (TG). The safety of ezetimibe in this subject population will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Each subject may be of either sex and of any race/ethnicity, and must be >=6 and <=10 years of age, with a diagnosis of primary hypercholesterolemia (heterozygous familial or nonfamilial) despite being on a lipid-lowering diet for at least 3 months with a LDL-C of >159mg/dL
* Each subject's parent/guardian must be willing to give written informed consent on his/her behalf.

Exclusion Criteria:

Each subject must not:

* Have known hypersensitivity or any contraindication to ezetimibe.
* Have use of any investigational drugs within 30 days of study entry.
* Be a member or a family member of the personnel of the investigational or sponsor staff directly involved with this trial.
* Be a female of child-bearing potential who is pregnant, intends to become pregnant, or is nursing
* Have known congenital cardiac disorder.
* Have documented or laboratory values consistent with homozygous familial hypercholesterolemia (HoFH).
* Be known to be human immunodeficiency virus (HIV) positive.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 138 (Actual)
Dates: Start 2009-05-21 (Actual); Primary Completion 2012-04-13 (Actual); Study Completion 2012-04-13 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kusters DM, Caceres M, Coll M, Cuffie C, Gagne C, Jacobson MS, Kwiterovich PO, Lee R, Lowe RS, Massaad R, McCrindle BW, Musliner TA, Triscari J, Kastelein JJ. Efficacy and safety of ezetimibe monotherapy in children with heterozygous familial or nonfamilial hypercholesterolemia. J Pediatr. 2015 Jun;166(6):1377-84.e1-3. doi: 10.1016/j.jpeds.2015.02.043. Epub 2015 Apr 1. PMID 25841542

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ezetimibe | Placebo
Started | 93 | 45
Completed | 89 | 45
Not Completed | 4 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetimibe | Placebo | Total
Number analyzed (Participants) | 93 | 45 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.2 (1.7) | 8.5 (1.6) | 8.3 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 27 | 79
  Male | 41 | 18 | 59

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) at Week 12
Description: Serum LDL-C levels calculated at baseline and after 12 weeks of study drug administration. LDL-C were calculated by the method of Friedewald equation, LDL-C = Total Cholesterol (TC) - (High-density lipoprotein cholesterol [HDL-C] + triglyceride [TG]/5).
Time Frame: Baseline and Week 12
Population: Full Analysis Set (FAS) population defined as all randomized participants who took at least one dose of study
  medication and had a baseline value and at least one valid post-baseline evaluation.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 85 | 42
Percent Change | -27.70 [-30.80 to -24.59] | -0.95 [-4.94 to 3.04]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -26.74, 95% CI 2-sided [-30.80 to -22.69]

2. Secondary Outcome: Percentage Change From Baseline in Total Cholesterol (TC) at Week 12
Description: Serum TC levels measured using enzymatic methods at baseline and after 12 weeks of study drug administration.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 85 | 42
Percentage Change | -20.74 [-23.29 to -18.18] | 0.19 [-3.07 to 3.44]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -20.92, 95% CI 2-sided [-24.20 to -17.65]

3. Secondary Outcome: Percentage Change From Baseline in Apolipoprotein B (Apo B) at Week 12
Description: Serum Apo B measured at baseline and after 12 weeks of study drug administration.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 85 | 42
Percent Change | -21.66 [-24.94 to -18.38] | -1.42 [-5.55 to 2.70]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -20.24, 95% CI 2-sided [-24.02 to -16.45]

4. Secondary Outcome: Percentage Change From Baseline High-density Lipoprotein Cholesterol (HDL-C) at Week 12
Description: Serum HDL-C levels measured by photometry after precipitation at baseline and after 12 weeks of study drug administration.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 85 | 42
Percentage Change | 2.11 [-2.27 to 6.48] | 1.41 [-4.14 to 6.96]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p = 0.807, ANCOVA; Difference in least-square means = 0.70, 95% CI 2-sided [-4.97 to 6.36]

5. Secondary Outcome: Percentage Change From Baseline in Non-HDL-C at Week 12
Description: Serum Non-HDL-C calculated at baseline and after 12 weeks of study drug administration. Non-HDL-C values were calculated as follows: Non-HDL-C (mg/dL) = TC - HDL-C.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 85 | 42
Percentage Change | -25.47 [-28.45 to -22.49] | 0.28 [-3.52 to 4.08]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Differrence in least-squares means = -25.75, 95% CI 2-sided [-29.59 to -21.91]

6. Secondary Outcome: Percentage Change From Baseline in Triglycerides (TG) at Week 12
Description: Serum TG levels measured using enzymatic methods at baseline and after 12 weeks of study drug.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 85 | 42
Percentage change | -6.23 [-12.73 to 0.75] | 8.44 [-2.03 to 20.03]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p = 0.021, Constrained longitudinal data analysis; Difference in least-square means = -14.68, 95% CI 2-sided [-27.35 to -2.00]

7. Secondary Outcome: Percent Change From Baseline in LDL-C at Week 2
Description: Serum LDL-C levels calculated at baseline and after 2 weeks of study drug administration. LDL-C were calculated by the method of Friedewald equation, LDL-C = Total Cholesterol (TC) - (High-density lipoprotein cholesterol [HDL-C] + triglyceride [TG]/5).
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 91 | 43
Percentage Change | -24.75 [-27.80 to -21.69] | 0.23 [-3.74 to 4.20]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -24.97, 95% CI 2-sided [-28.95 to -20.99]

8. Secondary Outcome: Percent Change From Baseline in LDL-C at Week 4
Description: Serum LDL-C levels calculated at baseline and after 4 weeks of study drug administration. LDL-C were calculated by the method of Friedewald equation, LDL-C = Total Cholesterol (TC) - (High-density lipoprotein cholesterol [HDL-C] + triglyceride [TG]/5).
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 90 | 43
Percentage Change | -26.93 [-29.81 to -24.05] | -2.99 [-6.66 to 0.68]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-square means = -23.94, 95% CI 2-sided [-27.49 to -20.39]

9. Secondary Outcome: Percent Change From Baseline in LDL-C at Week 8
Description: Serum LDL-C levels calculated at baseline and after 8 weeks of study drug administration. LDL-C were calculated by the method of Friedewald equation, LDL-C = Total Cholesterol (TC) - (High-density lipoprotein cholesterol [HDL-C] + triglyceride [TG]/5).
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 90 | 44
Percentage Change | -27.22 [-30.30 to -24.15] | 0.49 [-3.46 to 4.43]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -27.71, 95% CI 2-sided [-31.70 to -23.73]

10. Secondary Outcome: Percentage Change From Baseline in TC at Week 2
Description: Serum TC levels measured using enzymatic methods at baseline and after 2 weeks of study drug administration.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 91 | 43
Percentage Change | -18.69 [-21.21 to -16.18] | 1.40 [-1.83 to 4.63]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -20.09, 95% CI 2-sided [-23.30 to -16.89]

11. Secondary Outcome: Percentage Change From Baseline in TC at Week 4
Description: Serum TC levels measured using enzymatic methods at baseline and after 4 weeks of study drug administration.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 90 | 43
Percentage Change | -20.57 [-23.05 to -18.08] | -0.29 [-3.45 to 2.86]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -20.27, 95% CI 2-sided [-23.39 to -17.15]

12. Secondary Outcome: Percentage Change From Baseline in TC at Week 8
Description: Serum TC levels measured using enzymatic methods at baseline and after 8 weeks of study drug administration.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 90 | 44
Percentage Change | -20.84 [-23.40 to -18.27] | 0.54 [-2.73 to 3.81]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -21.37, 95% CI 2-sided [-24.67 to -18.08]

13. Secondary Outcome: Percentage Change From Baseline HDL-C at Week 2
Description: Serum HDL-C levels measured by photometry after precipitation at baseline and after 2 weeks of study drug administration.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 91 | 43
Percentage Change | 0.01 [-4.28 to 4.30] | 0.96 [-4.51 to 6.43]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p = 0.733, ANCOVA; Difference in least-squares means = -0.95, 95% CI 2-sided [-6.46 to 4.55]

14. Secondary Outcome: Percentage Change From Baseline HDL-C at Week 4
Description: Serum HDL-C levels measured by photometry after precipitation at baseline and after 4 weeks of study drug administration.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 90 | 43
Percentage Change | 0.86 [-3.69 to 5.42] | 0.33 [-5.54 to 6.19]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p = 0.863, ANCOVA; Difference in least-squares means = 0.53, 95% CI 2-sided [-5.59 to 6.66]

15. Secondary Outcome: Percentage Change From Baseline HDL-C at Week 8
Description: Serum HDL-C levels measured by photometry after precipitation at baseline and after 8 weeks of study drug administration.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 90 | 44
Percentage Change | 1.41 [-2.95 to 5.77] | -0.52 [-6.04 to 5.00]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p = 0.501, ANCOVA; Difference in least-squares means = 1.92, 95% CI 2-sided [-3.71 to 7.56]

16. Secondary Outcome: Percentage Change From Baseline in Non-HDL-C at Week 2
Description: Serum Non-HDL-C calculated at baseline and after 2 weeks of study drug administration. Non-HDL-C values were calculated as follows: Non-HDL-C (mg/dL) = TC - HDL-C.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 91 | 43
Percentage Change | -22.54 [-25.41 to -19.67] | 1.64 [-2.03 to 5.30]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -24.18, 95% CI 2-sided [-27.78 to -20.58]

17. Secondary Outcome: Percentage Change From Baseline in Non-HDL-C at Week 4
Description: Serum Non-HDL-C calculated at baseline and after 4 weeks of study drug administration. Non-HDL-C values were calculated as follows: Non-HDL-C (mg/dL) = TC - HDL-C.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 90 | 43
Percentage Change | -24.94 [-27.75 to -22.14] | -0.33 [-3.88 to 3.22]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -24.61, 95% CI 2-sided [-28.06 to -21.16]

18. Secondary Outcome: Percentage Change From Baseline in Non-HDL-C at Week 8
Description: Serum Non-HDL-C calculated at baseline and after 8 weeks of study drug administration. Non-HDL-C values were calculated as follows: Non-HDL-C (mg/dL) = TC - HDL-C.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 90 | 44
Percentage Change | -25.41 [-28.37 to -22.45] | 1.14 [-2.63 to 4.92]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -26.55, 95% CI 2-sided [-30.35 to -22.75]

19. Secondary Outcome: Percentage Change From Baseline in TG at Week 2
Description: Serum TG levels measured using enzymatic methods at baseline and after 2 weeks of study drug administration.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 91 | 43
Percentage Change | -3.90 [-10.66 to 3.37] | 5.83 [-4.76 to 17.59]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p = 0.137, Constrained longitudinal data analysis; Difference in least-squares means = -9.73, 95% CI 2-sided [-22.73 to 3.27]

20. Secondary Outcome: Percentage Change From Baseline in TG at Week 4
Description: Serum TG levels measured using enzymatic methods at baseline and after 4 weeks of study drug administration.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 90 | 43
Percentage Change | -5.54 [-11.05 to 0.31] | 9.65 [0.60 to 19.53]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p = 0.005, Constrained longitudinal data analysis; Difference in least-squares means = -15.19, 95% CI 2-sided [-26.05 to -4.34]

21. Secondary Outcome: Percentage Change From Baseline in TG at Week 8
Description: Serum TG levels measured using enzymatic methods at baseline and after 8 weeks of study drug administration.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 90 | 44
Percentage Change | -9.99 [-16.28 to -3.21] | -1.38 [-11.02 to 9.31]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p = 0.149, Constrained longitudinal data analysis; Difference in least-squares means = -8.61, 95% CI 2-sided [-20.44 to 3.23]

22. Secondary Outcome: Percentage Change From Baseline in Apolipoprotein A-I (Apo A-I) at Week 12
Description: Serum Apo A-I levels measured at baseline and after 12 weeks of study drug administration.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 85 | 42
Percentage Change | 1.80 [-1.86 to 5.46] | 3.71 [-0.87 to 8.30]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p = 0.373, ANCOVA; Difference in least-squares means = -1.91, 95% CI 2-sided [-6.15 to 2.32]

23. Secondary Outcome: Percentage Change From Baseline in TC:HDL-C Ratio at Week 2
Description: Serum TC:HDL-C Ratio calculated at baseline and after 2 weeks of study drug administration.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 91 | 43
Percentage Change | -17.21 [-21.08 to -13.34] | 2.56 [-2.37 to 7.48]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in Least-squares mean = -19.76, 95% CI 2-sided [-24.70 to -14.82]

24. Secondary Outcome: Percentage Change From Baseline in TC:HDL-C Ratio at Week 4
Description: Serum TC:HDL-C Ratio calculated at baseline and after 4 weeks of study drug administration.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 90 | 43
Percentage Change | -19.36 [-23.16 to -15.56] | 1.48 [-3.30 to 6.25]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -20.83, 95% CI 2-sided [-25.59 to -16.07]

25. Secondary Outcome: Percentage Change From Baseline in TC:HDL-C Ratio at Week 8
Description: Serum TC:HDL-C Ratio calculated at baseline and after 8 weeks of study drug administration.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 90 | 44
Percentage Change | -20.07 [-24.20 to -15.94] | 3.41 [-1.87 to 8.70]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -23.48, 95% CI 2-sided [-29.00 to -17.97]

26. Secondary Outcome: Percentage Change From Baseline in TC:HDL-C Ratio at Week 12
Description: Serum TC:HDL-C Ratio calculated at baseline and after 12 weeks of study drug administration.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 85 | 42
Percentage Change | -21.09 [-24.98 to -17.19] | 1.20 [-3.70 to 6.11]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -22.29, 95% CI 2-sided [-27.25 to -17.34]

27. Secondary Outcome: Percentage Change From Baseline in LDL-C:HDL-C Ratio at Week 2
Description: Serum LDL-C:HDL-C Ratio calculated at baseline and after 2 weeks of study drug administration.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 91 | 43
Percentage Change | -23.35 [-27.69 to -19.01] | 1.15 [-4.35 to 6.65]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -24.50, 95% CI 2-sided [-29.88 to -19.12]

28. Secondary Outcome: Percentage Change From Baseline in LDL-C:HDL-C Ratio at Week 4
Description: Serum LDL-C:HDL-C Ratio calculated at baseline and after 4 weeks of study drug administration.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 90 | 42
Percentage Change | -25.72 [-30.12 to -21.33] | -0.57 [-6.14 to 5.00]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -25.15, 95% CI 2-sided [-30.69 to -19.62]

29. Secondary Outcome: Percentage Change From Baseline in LDL-C:HDL-C Ratio at Week 8
Description: Serum LDL-C:HDL-C Ratio calculated at baseline and after 8 weeks of study drug administration.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 90 | 43
Percentage Change | -26.43 [-31.21 to -21.66] | 2.87 [-3.28 to 9.02]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -29.31, 95% CI 2-sided [-35.71 to -22.91]

30. Secondary Outcome: Percentage Change From Baseline in LDL-C:HDL-C Ratio at Week 12
Description: Serum LDL-C:HDL-C Ratio calculated at baseline and after 12 weeks of study drug administration.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 85 | 42
Percentage Change | -28.01 [-32.65 to -23.36] | 0.34 [-5.57 to 6.25]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -28.35, 95% CI 2-sided [-34.41 to -22.29]

31. Secondary Outcome: Percentage Change From Baseline in Apo B:Apo A-I Ratio at Week 12
Description: Serum Apo B:Apo A-I Ratio calculated at baseline and after 12 weeks of study drug administration
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 85 | 42
Percentage Change | -22.16 [-26.13 to -18.19] | -2.87 [-7.84 to 2.09]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -19.28, 95% CI 2-sided [-23.87 to -14.70]

32. Secondary Outcome: Percentage Change From Baseline in High-sensitivity C-reactive Protein (Hs-CRP) at Week 4
Description: Plasma hs-CRP measured at baseline and after 4 weeks of study drug administration.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 90 | 43
Percentage Change | 10.00 [-15.65 to 43.45] | 56.11 [7.68 to 126.32]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p = 0.116, Constrained longitudinal data analysis; Difference in least-squares means = -46.11, 95% CI 2-sided [-108.14 to 15.92]

33. Secondary Outcome: Percentage Change From Baseline in High-sensitivity C-reactive Protein (Hs-CRP) at Week 12
Description: Plasma hs-CRP measured at baseline and after 12 weeks of study drug administration.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 85 | 42
Percentage Change | 9.35 [-13.47 to 38.19] | -7.92 [-33.48 to 27.46]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p = 0.382, Constrained longitudinal data analysis; Difference in least-squares means = 17.27, 95% CI 2-sided [-20.46 to 55.00]

34. Secondary Outcome: Percent Change From Baseline in Sitosterol at Week 2
Description: Plasma sitosterol measured at baseline and after 2 weeks of study drug administration.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 89 | 43
Percentage Change | -50.20 [-54.65 to -45.76] | -0.59 [-6.26 to 5.08]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -49.61, 95% CI 2-sided [-55.36 to -43.87]

35. Secondary Outcome: Percentage Change From Baseline in Sitosterol at Week 4
Description: Plasma sitosterol measured at baseline and after 4 weeks of study drug administration.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 87 | 43
Percentage Change | -58.82 [-63.04 to -54.61] | -0.30 [-5.52 to 4.93]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -58.52, 95% CI 2-sided [-63.67 to -53.38]

36. Secondary Outcome: Percentage Change From Baseline in Sitosterol at Week 8
Description: Plasma sitosterol measured at baseline and after 8 weeks of study drug administration.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 86 | 44
Percentage Change | -61.59 [-66.39 to -56.78] | -0.57 [-6.69 to 5.56]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -61.02, 95% CI 2-sided [-67.51 to -54.53]

37. Secondary Outcome: Percentage Change From Baseline in Sitosterol at Week 12
Description: Plasma sitosterol measured at baseline and after 12 weeks of study drug administration.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 82 | 41
Percentage Change | -60.65 [-67.39 to -53.92] | 2.09 [-7.01 to 11.18]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA; Difference in least-squares means = -62.74, 95% CI 2-sided [-73.22 to -52.26]

38. Secondary Outcome: Percentage Change From Baseline in Campesterol at Week 2
Description: Plasma campesterol measured at baseline and after 2 weeks of study drug administration.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 89 | 43
Percentage Change | -53.87 [-57.99 to -49.74] | -4.38 [-9.66 to 0.90]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -49.48, 95% CI 2-sided [-54.83 to -44.14]

39. Secondary Outcome: Percentage Change From Baseline in Campesterol at Week 4
Description: Plasma campesterol measured at baseline and after 4 weeks of study drug administration.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 87 | 43
Percentage Change | -62.27 [-66.21 to -58.32] | -4.28 [-9.20 to 0.65]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -57.99, 95% CI 2-sided [-62.87 to -53.11]

40. Secondary Outcome: Percentage Change From Baseline in Campesterol at Week 8
Description: Plasma campesterol measured at baseline and after 8 weeks of study drug administration.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 86 | 44
Percentage Change | -66.79 [-71.21 to -62.37] | -4.19 [-9.83 to 1.45]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -62.60, 95% CI 2-sided [-68.54 to -56.66]

41. Secondary Outcome: Percentage Change From Baseline in Campesterol at Week 12
Description: Plasma campesterol measured at baseline and after 12 weeks of study drug administration.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 82 | 41
Percentage Change | -67.59 [-73.68 to -61.50] | -2.92 [-11.15 to 5.31]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -64.67, 95% CI 2-sided [-74.11 to -55.23]

42. Secondary Outcome: Percentage Change From Baseline in Cholestanol at Week 2
Description: Plasma cholestanol measured at baseline and after 2 weeks of study drug administration.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 89 | 43
Percentage Change | -25.44 [-30.30 to -20.59] | -7.09 [-13.29 to -0.90]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -18.35, 95% CI 2-sided [-24.70 to -11.99]

43. Secondary Outcome: Percentage Change From Baseline in Cholestanol at Week 4
Description: Plasma cholestanol measured at baseline and after 4 weeks of study drug administration.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 87 | 43
Percentage Change | -27.40 [-31.95 to -22.85] | -1.79 [-7.42 to 3.85]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -25.61, 95% CI 2-sided [-31.20 to -20.02]

44. Secondary Outcome: Percentage Change From Baseline in Cholestanol at Week 8
Description: Plasma cholestanol measured at baseline and after 8 weeks of study drug administration.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 86 | 44
Percentage Change | -29.19 [-33.98 to -24.39] | -0.44 [-6.44 to 5.56]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -28.74, 95% CI 2-sided [-34.89 to -22.59]

45. Secondary Outcome: Percentage Change From Baseline in Cholestanol at Week 12
Description: Plasma cholestanol measured at baseline and after 12 weeks of study drug administration.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 82 | 41
Percentage Change | -28.71 [-34.44 to -22.99] | 3.42 [-4.07 to 10.92]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = -32.14, 95% CI 2-sided [-40.38 to -23.90]

46. Secondary Outcome: Percentage Change From Baseline in Lathosterol at Week 2
Description: Plasma lathosterol measured at baseline and after 2 weeks of study drug administration.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 89 | 43
Percentage Change | 34.07 [24.68 to 43.45] | 14.06 [2.22 to 25.90]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA; Difference in least-squares means = 20.01, 95% CI 2-sided [8.10 to 31.91]

47. Secondary Outcome: Percentage Change From Baseline in Lathosterol at Week 4
Description: Plasma lathosterol measured at baseline and after 4 weeks of study drug administration.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 87 | 43
Percentage Change | 33.02 [23.44 to 42.60] | 6.73 [-5.27 to 18.73]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = 26.29, 95% CI 2-sided [13.99 to 38.58]

48. Secondary Outcome: Percentage Change From Baseline in Lathosterol at Week 8
Description: Plasma lathosterol measured at baseline and after 8 weeks of study drug administration.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 86 | 44
Percentage Change | 35.87 [26.14 to 45.61] | -0.82 [-12.99 to 11.34]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = 36.70, 95% CI 2-sided [24.12 to 49.28]

49. Secondary Outcome: Percentage Change From Baseline in Lathosterol at Week 12
Description: Plasma lathosterol measured at baseline and after 12 weeks of study drug administration.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 82 | 41
Percentage Change | 36.62 [26.46 to 46.78] | 12.57 [-0.36 to 25.50]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least-squares means = 24.05, 95% CI 2-sided [10.43 to 37.67]

ADVERSE EVENTS:
Description: Safety analysis was performed on the All-Patients-as-Treated (APaT) Population defined as all randomized patients who received at least one dose of double-blind study therapy.
Arm/Group | Ezetimibe | Placebo
Serious Adverse Events (participants affected / at risk) | 2/92 | 0/45
Other Adverse Events (participants affected / at risk) | 27/92 | 18/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe (N=92) | Placebo (N=45)
Epilepsy congenital (Congenital, familial and genetic disorders) | 1 (3) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe (N=92) | Placebo (N=45)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 4 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3)
Influenza (Infections and infestations) | 5 (5) | 3 (3)
Nasopharyngitis (Infections and infestations) | 10 (10) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 1 (1)
Headache (Nervous system disorders) | 4 (9) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agreed not to publish or publicly present any interim results of the trial without the prior written consent of the sponsor. The investigator further agreed to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial.